CLINICAL TRIAL: NCT04394026
Title: COVID-19 Imaging Features
Brief Title: Imaging Feature of SARS-CoV2 Infection
Acronym: COVID19IF
Status: Completed | Type: Observational
Sponsor: Francesco De Cobelli (Other)
Responsible Party: Sponsor-Investigator, Francesco De Cobelli, MD, Chair Radiology Department, IRCCS San Raffaele
Organization: IRCCS San Raffaele (Other)
Other Study IDs: COVID-19 IF
Record Dates: First submitted 2020-05-15; First posted 2020-05-19 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Viral Pneumonia; COVID
Keywords: diagnosis; disease progression; imaging features; SARS-CoV2; COVID
MeSH Terms: conditions — Pneumonia, Viral; Disease; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The novel coronavirus SARS-CoV2 clinically presents with pneumonia, characterised by fever, cough, dyspnea. The severity of the disease varies widely with evidence of mild disease in the majority of confirmed cases, severe pneumonia-dyspnea, hypoxia or lung involvement at imaging within 24-48 hours- and critical disease with respiratory failure, shock or multi-organ failure in particular patient cohorts. Imaging plays a key role is diagnosis and progression of this disease.

DETAILED DESCRIPTION:
In March 2020, the third highest number of positive cases in the world was recorded in Italy, mainly due to 2 outbreaks of 2 different clusters in Lombardy and Veneto.

Fever is the most common symptom, followed by fatigue and dry cough; worsening of dyspnea and acute respiratory distress syndrome are found in severe cases. Previous reports have highlighted the key role of chest computed tomography (CT) and chest X-ray (CXR) in the diagnosis and follow-up of CoViD-19.

The most frequent clinical manifestation seems to be viral pneumonia, characterised by fever, cough, dyspnea. The severity of the disease varies widely: with evidence of mild disease in the majority of confirmed cases, severe pneumonia on a part of these, defined as dyspnea, hypoxia or lung involvement > 40% at imaging within 24-48 hours, and critical disease defined as respiratory failure, shock or multi-organ failure in particular patient cohorts.The mortality rate between cases ranges from approximately 4% in early reports to 14%, depending on the intensity of transmission and time of infection, and most fatal cases occurred in older patients or in patients with pre-existing medical co-morbidities.

Imaging plays an essential role in the diagnosis and follow-up of this infection.Several studies have been published describing the results of imaging, mainly using chest CT (computed tomography) with a limited number of articles describing disease in European patients or the possible different clinical/radiological presentation of the disease in European patients.

Pulmonary pathological findings appear to be similar to those previously described in SARS and MERS, with a prevalence of frosted glass densities and occasional consolidation.According to the literature, the 3 main features for the diagnosis of CoVid-19 pneumonia are: alveolar disease, represented by ground glass densities, bilateral distribution and prevalent peripheral involvement. This triad is more common in intermediate stages of the disease. In the early stages of the disease, a significant proportion of patients may present with negative or dubious X-rays and CT scans.There is an important overlap with imaging findings of other viral pneumonia, in particular with other members of the coronaviridae family: consolidation, however, seems to be less common in the early stages of CoViD-19 and bilateral distribution is less frequent in SARS and MERS pneumonia. Very little data have been published on the radiological evolution and modification of radiological aspects during infection: as the disease progresses, parenchymal consolidations begin to resorb and assume a frosted glass appearance. Another possible evolution is the progression towards the radiological aspect of the "white lung". This study aims to describe imaging aspects of CoViD-19 infection in Italian patients and the data on the radiological evolution.

ELIGIBILITY:
Inclusion Criteria:

* CoViD-19 positive patients (rRT-PCR naso-pharyngeal swab)
* Suspicion of SARS-CoV2 on chest X-ray and/or chest CT presentation of disease
* Patients of all ages
* Subjects at risk (minors, patients in emergency situations, pregnant women, potentially incapable of giving their consent )
* Having signed the Informed Consent

Exclusion Criteria:

* Not fulfilling any of the above

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with proven COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-04-16 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Describe qualitative and quantitative variables | Through study completion, an average of 5 months
  Evaluate RX imaging aspects at the time of diagnosis and until discharge.
Describe qualitative and quantitative variables | Through study completion, an average of 5 months
  Evaluate CT imaging aspects at the time of diagnosis and until discharge.
Ability of imaging to predict disease progression | Through study completion, an average of 5 months
  Correlate imaging findings to OS
Ability of imaging to predict disease evolution | Through study completion, an average of 5 months
  Correlate imaging findings over time

SECONDARY OUTCOMES:
Imaging findings and demographic data | Through study completion, an average of 5 months
  Correlate imaging findings to age and sex
Imaging findings and laboratory exams | Through study completion, an average of 5 months
  Correlate imaging findings to laboratory values

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Martinenghi, MD, Principal Investigator — IRCCS Ospedale San Raffaele
Locations (1):
- Deaprtment of Radiology, IRCCS Ospedale San Raffaele, Milan, Italy